CLINICAL TRIAL: NCT03951454
Title: Taking Time to Connect: A Randomized Clinical Trial for Hispanic Mothers Diagnosed With Cancer
Brief Title: Taking Time to Connect: A Study of Programs for Hispanic Mothers Diagnosed With Cancer and Their Children
Acronym: TTTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico State University (Other)
Collaborators: University of Washington (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Rebecca Palacios, Associate Professor, New Mexico State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17894
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Cancer Survivorship
Keywords: maternal; non-metastatic; anxiety; depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Experimental group: Experimental subjects will receive Conexiones, a program designed to help the cancer-diagnosed mother manage her child's cancer-related concerns by improving the mother's mood and anxiety and by equipping the mother with parenting and communication skills to assist the child in coping with the mother's cancer. The program involves 5 fully scripted telephone-delivered educational sessions delivered at 2-week intervals by patient educators.
  Control group: Control subjects will receive an informational booklet published by NCI called, "Taking Time." The booklet contains information on ways to manage emotional issues, including the importance of sharing feelings about the cancer with a trusted adult confidant, learning all you can about your cancer in order to regain control and talking with medical providers, and dealing with a new self-image. This group receives one scripted telephone-delivered session guiding the mother on how to obtain the most from the booklet.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are not informed as to whether they are in the experimental intervention or the control intervention.
  Members of the Data Collection Team at New Mexico State University (NMSU) remain "blind" on the randomization status of study participants. Randomization will be handled centrally by the team's biostatistician, Griffith, at the University of Washington. She will be responsible for centralized random assignment using block randomization [by recruitment sites, language of program delivery, and cancer types] and will communicate that assignment only to Palacios, Lewis and the Project Manager.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conexiones (Experimental): 5 telephone sessions of Conexiones, with each session delivered 2 weeks apart across a total period of 8 weeks
  Interventions: Behavioral: Conexiones
- Taking Time (Other): 1 telephone session consisting of a scripted protocol guiding participants through the NCI's Taking Time Booklet.
  Interventions: Behavioral: Taking Time

INTERVENTIONS:
Behavioral: Conexiones — 5 Conexiones telephone sessions
  Arms: Conexiones
Behavioral: Taking Time — 1 Taking Time telephone session
  Arms: Taking Time

SUMMARY:
This NCI-funded randomized clinical trial (RCT) will test the short-term efficacy of Conexiones, a culturally adapted cancer education program designed to help Hispanic mothers diagnosed with cancer and their children to cope with cancer.

DETAILED DESCRIPTION:
The purpose of the proposed study is to test the short-term efficacy of a cancer parenting education program for diagnosed child-rearing Hispanic mothers, called Conexiones. This program was culturally adapted from a parenting program previously tested for efficacy in a Phase III, 6-state randomized clinical trial. However, the original program was tested on primarily non-Hispanic White (NHW) mothers with breast cancer. The Conexiones program represents a culturally adapted version of the original parenting program and is now ready for testing with Hispanic mothers living in the Border States of New Mexico and Texas. Eligible women will be diagnosed within the last 2 years with a primary, non-advanced cancer (stages 0-III) of any type and will be mothers of a child 5-17 years of age. Study participants will be recruited from medical providers, local channels (e.g. community health agencies, Community Health Worker networks, social media), and through self-referral in the recruitment counties. After completing signed informed consent and baseline measures, mothers will be randomized to an experimental or control group. All program materials/delivery are available in English and Spanish. All program education and data collection is conducted entirely by telephone so that the women can participate within the comfort of their homes and at times convenient for them. The experimental group will receive 5 fully scripted telephone-delivered educational sessions every 2 weeks by specially trained patient educators. The control group will receive "Taking Time," a NCI cancer education booklet, and 1 scripted telephone-delivered session with a patient educator. Assessments will occur at 3 months post-baseline for all participants and at 6 months post-baseline for 66% of participants. Post-intervention measures consist of standardized questionnaires with well-established validity and reliability, all available in Spanish. Linear Mixed Models will be used to analyze outcomes within an intent to treat analysis.. With an estimated Effect size of 0.52 for the primary outcome measure of the child's behavioral-emotional adjustment, the investigators need to retain a total sample size of 116 (58/group) for efficacy analysis. The investigators plan to enroll 156 eligible mothers, allowing for an expected 25% attrition rate from all causes. Study results will be essential as a next step in testing Conexiones with other Hispanic subgroups in a larger trial and readying the program for wider testing and dissemination to provider and non-profit organizations serving Hispanic parents with cancer throughout the United States.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic women
* Diagnosed with primary, non-metastatic cancer (stage 0, I, II, or III) of any type in the past 2 years
* Has a child 5 to 17 years old living at home and who knows about their mother's cancer
* Lives in New Mexico or Texas
* Has ready access to a telephone
* Can read and write in English or Spanish

Exclusion Criteria:

* Has a secondary and/or recurrent cancer diagnosis
* Diagnosed with basal or squamous cell carcinoma
* Not able to read or write in English or Spanish
* Does not have ready access to a telephone
* Her child is not aware of the mother's cancer diagnosis
* Her child has learning challenges that would prevent him/her from engaging in a conversation with their mother

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only mothers diagnosed with cancer may participate in the trial.
Enrollment: 43 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Child Behavior Checklist (CBCL) | 3 months
  A mother-reported scale of a broad range of behavior problems in children ages 6-18; Response options range from 0 to 2 from "Not True (as far as you know)" to "Somewhat or Sometimes True" to "Very True or Often True

SECONDARY OUTCOMES:
Center for Epidemiological Studies-Depression Scale (CES-D) | 7 days
  Measures maternal depressed mood; 15 items measured on a 4 point Likert-type scale (1 -Rarely or none of the time; 4-Most or all of the time)
Spielberger State-Trait Anxiety Inventory (STAI) | 1 hour
  Measures maternal anxiety; 20 items; 4 point Likert-type scale (1-Not at all; 4-Very much so)
Cancer Self-Efficacy Scale (CASE) | 1 hour
  Three subscales (Help Child, Deal & Manage, and Stay Calm) measure parenting self-efficacy; 28 items; 11 point Likert-type scale (0-not at all confident; 10-Very Confident)
Family-Peer Relationship Scale (FPRQ) | 3 months
  Measures parenting quality using 7 items that assess interpersonal communication between the mother and child; includes 2 subscales (Disclosure of Negative Feelings and Disclosure of Bad Things Happening); 5 point Likert-type scale (0-Never talks about it; 4-Always talks about it)
Parenting Skills Checklist | 1 hour
  Assesses the interactional behaviors mothers used to assist their child to disclose, discuss, and cope with the breast cancer; 2 subscales (Elicitation subscale, Connecting & Coping subscale); 8 items; 6 point Likert-type scale (0-Never; 5-All of the time)

OTHER OUTCOMES:
Social Support Survey Instrument | 3 months
  Assesses emotional and informational support, 9 items; 5 point Likert type scale (0-none of the time; 4-all of the time)
Brief Cope | 3 months
  Measure of strategies used for coping or regulating cognitions in response to stressors; 28 items; 4 point Likert type scale (1-I didn't do this at all; 4-I did this a lot)
COVID-19 Impact of the Pandemic in Cancer Patients and Survivors: Psychosocial & Practical Experiences- COVID-19 Specific Distress Subscale | 1 hour
  13 items assessing COVID 19 specific distress among cancer patients/survivors; participants respond on a 5 point Likert type scale (1-Strongly Disagree; 5- Strongly Agree)
COVID-19 Impact of the Pandemic in Cancer Patients and Survivors: Psychosocial & Practical Experiences - Health Care Disruptions & Concerns Subscale | 1 hour
  4 items assess COVID-19 related health care disruptions and concerns among cancer patients/survivors; participants respond on a 5 point Likert type scale (1-Strongly Disagree; 5- Strongly Agree)
COVID-19 Impact of the Pandemic in Cancer Patients and Survivors: Psychosocial & Practical Experiences - Disruption to Daily Activities & Social Interactions Subscale | 1 hour
  6 items assess COVID-19 related disruption to daily activities & social interactions among cancer patients/survivors; participants respond on a 5 point Likert type scale (1-Strongly Disagree; 5- Strongly Agree)
COVID-19 Impact of the Pandemic in Cancer Patients and Survivors: Psychosocial & Practical Experiences- Financial Hardship Subscale | 1 hour
  5 items assess COVID-19 related financial hardships among cancer patients/survivors; participants respond on a 5 point Likert type scale (1-Strongly Disagree; 5- Strongly Agree)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Palacios, PhD, Principal Investigator — New Mexico State University; Frances M Lewis, PhD, Principal Investigator — University of Washington, Fred Hutchinson Cancer Research Center
Locations (5):
- United States (5):
  - New Mexico State University, Las Cruces, New Mexico
  - Memorial Medical Center-Cancer Center, Las Cruces, New Mexico
  - The Hospitals of Providence, El Paso, Texas
  - University Medical Center of El Paso, El Paso, Texas
  - Mays Cancer Center, UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data obtained on all standardized measures at baseline and post intervention will be shared with investigators both internal and external to New Mexico State University, the University of Washington, and the Fred Hutchinson Cancer Research Center. Prior to sharing the data, Lewis (Co-PI) and Palacios (Co-PI) will request a detailed plan for data analysis, the choice of the study sample, and a rationale and significance for the proposal. Prior to releasing the data, the proposal will be reviewed by Lewis and Palacios. Access levels will be set to protect subject identification and unique identifiers linked to participant identity will be stripped, (i.e., data will be de-identified). Access will be made available as soon as the primary analyses are completed and accepted for publication in a professional journal and secondary analyses are completed by the team's investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Access will be made available as soon as the primary analyses are completed and accepted for publication in a professional journal and secondary analyses are completed by the team's investigators.
Access Criteria: Prior to sharing the data, Lewis (Co-PI) and Palacios (Co-PI) will request a detailed plan for data analysis, the choice of the study sample, and a rationale and significance for the proposal. Prior to releasing the data, the proposal will be reviewed by Lewis and Palacios.

REFERENCES:
- [Background] Lewis FM, Casey SM, Brandt PA, Shands ME, Zahlis EH. The enhancing connections program: pilot study of a cognitive-behavioral intervention for mothers and children affected by breast cancer. Psychooncology. 2006 Jun;15(6):486-97. doi: 10.1002/pon.979. PMID 16216035
- See also: Complementary and Alternative Medicine Questionnaire — https://healthpolicy.ucla.edu/chis/design/Documents/CHIS2001_chiscam_q.pdf
- See also: Child Behavior Checklist for Ages 6-18 — https://aseba.org/wp-content/uploads/2019/02/schoolagecbcl.pdf
- See also: Brief COPE Inventory — https://scienceofbehaviorchange.org/measures/brief-cope/
- See also: COVID-19: Impact of the Pandemic and HRQoL in Cancer Patients and Survivors (IPHCPS) — https://www.phenxtoolkit.org/toolkit_content/PDF/UMiami_HRQoL.pdf